CLINICAL TRIAL: NCT03971136
Title: Evaluation of the Interest of Pulmonary Ultrasound in the Diagnosis and Early Detection of Acute Thoracic Syndrome in Hospitalized Children for Vaso-occlusive Sickle Cell Crisis: Multicenter Prospective Study
Brief Title: Pulmonary Ultrasound in the Diagnosis of Acute Thoracic Syndrome in Vaso-occlusive Sickle Cell Crisis
Acronym: ECHO-STA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ECHO-STA
Record Dates: First submitted 2019-05-23; First posted 2019-06-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Sickle-Cell Disease Nos With Crisis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with sickle cell disease (Other): Child from 12 months to 18 years old admitted for vaso-occlusive crisis
  Interventions: Diagnostic Test: pulmonary ultrasound

INTERVENTIONS:
Diagnostic Test: pulmonary ultrasound — The subjects will have an ultrasound on admission and on day 1, 2 and 3

SUMMARY:
ATS (acute thoracic syndrome) refers to acute pulmonary involvement in a sickle cell patient. The diagnosis is based on the association of clinical signs (fever or respiratory symptoms) with a recent pulmonary infiltrate on the chest x-ray.

The main objective of the study is to evaluate the place of the pulmonary ultrasound for the diagnosis of ATS, in comparison with frontal chest x-ray.

DETAILED DESCRIPTION:
The ATS occurs in half of the cases during hospitalization for a VOC (Vaso Occlusive crisis). The morbidity of ATS is important (respiratory insufficiency, duration of hospitalization, stays in intensive care, brain complications, pain, hypoxia, long-term sequelae, etc.) but no study has shown the benefits of curative treatments such as transfusion ( recommended at the time of diagnosis and practiced by some teams) or noninvasive ventilation (practiced by other teams). The first step before studying curative treatments is to have tools for early detection of ATS. Recent studies show non-inferiority of pulmonary ultrasonography compared to radiography and thoracic computed tomography in the diagnosis of pulmonary condensation (in adults and children). In a study performed in sickle cell adults admitted for ATS, pulmonary ultrasound was more sensitive than X-ray in detecting images of pulmonary consolidations visible on the chest CT scan.

Daswani et al have also shown the value of pulmonary ultrasound in comparison with radiography in the detection of consolidation lesions, suggestive of STA, in febrile children or young adults with sickle cell disease. They showed a good sensitivity (87%) and specificity (94%) of the pulmonary ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥12 months and <18 years
* Has a major sickle cell disease whatever the genotype
* Admission to hospital for a febrile vaso-occlusive crisis (VOC) or not
* Evolving at home for less than 48h
* Concomitant treatment with hydroxycarbamide / hydroxyurea possible
* Signed consent
* Patients affiliated to a French social security scheme

Exclusion Criteria:

* Child presenting an acute thoracic syndrome (ATS) from the outset at the admission
* Child who presented an ATS in the month preceding the inclusion
* Child in regular transfusion program or child who has received a hematopoietic stem cell transplant
* Child hospitalized at least 5 times for VOC in the year preceding inclusion (psychic problems making difficult the evaluation of the pain)
* Child who has already been included in the study during a previous VOC (each child participates in the study only once)
* VOC evolving for more than 48 hours before admission to the emergency room
* Acute splenic sequestration crisis at admission

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of pulmonary ultrasound | Day 1
  Proportion of subjects with positive pulmonary ultrasound among those with a positive chest X-ray at time t with 95% confidence interval at day 1
Sensitivity of pulmonary ultrasound | Day 2
  Proportion of subjects with positive pulmonary ultrasound among those with a positive chest X-ray at time t with 95% confidence interval at day 2
Sensitivity of pulmonary ultrasound | Day 3
  Proportion of subjects with positive pulmonary ultrasound among those with a positive chest X-ray at time t with 95% confidence interval at day 3

SECONDARY OUTCOMES:
Specificity of pulmonary ultrasound | Day 1
  Proportion of subjects with a positive pulmonary ultrasound among those with a negative chest X-ray at time t at day 1
Specificity of pulmonary ultrasound | Day 2
  Proportion of subjects with a positive pulmonary ultrasound among those with a negative chest X-ray at time t at day 2
Specificity of pulmonary ultrasound | Day 3
  Proportion of subjects with a positive pulmonary ultrasound among those with a negative chest X-ray at time t at day 3
Sensitivity of pulmonary ultrasound in relation with ATS diagnosis | day -3 of ATS diagnosis
  Proportion of subjects with positive pulmonary ultrasound among those with a positive chest X-ray at time t with 95% confidence intervalat day -3 of ATS diagnosis
Sensitivity of pulmonary ultrasound in relation with ATS diagnosis | day -1 of ATS diagnosis
  Proportion of subjects with positive pulmonary ultrasound among those with a positive chest X-ray at time t with 95% confidence interval at day -1 of ATS diagnosis
Sensitivity of pulmonary ultrasound in relation with ATS diagnosis | day -2 of ATS diagnosis
  Proportion of subjects with positive pulmonary ultrasound among those with a positive chest X-ray at time t with 95% confidence interval at day -2 of ATS diagnosis
Specificity of pulmonary ultrasound in relation with ATS diagnosis | day -1 of ATS diagnosis
  Proportion of subjects with a positive pulmonary ultrasound among those with a negative chest X-ray at time t at day -1 of ATS diagnosis
Specificity of pulmonary ultrasound in relation with ATS diagnosis | -3 day of ATS diagnosis
  Proportion of subjects with a positive pulmonary ultrasound among those with a negative chest X-ray at time t at day -3 of ATS diagnosis
Specificity of pulmonary ultrasound in relation with ATS diagnosis | day -2 of ATS diagnosis
  Proportion of subjects with a positive pulmonary ultrasound among those with a negative chest X-ray at time t at day -2 of ATS diagnosis

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital Antoine Béclère, Clamart
  - Centre Hospitalier Intercommunal Créteil, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Armand Trousseau, Paris

IPD SHARING:
Plan to Share IPD: No